CLINICAL TRIAL: NCT03844308
Title: Guided Meditation as a Wellness Tool in Anesthesia Providers
Brief Title: Wellness Tool in Anesthesia Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Associate Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2018P000387
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Burnout, Professional; Occupational Stress; Affective Symptoms
MeSH Terms: conditions — Burnout, Professional; Occupational Stress; Affective Symptoms

STUDY DESIGN:
Intervention Model Description: It is a waitlisted controlled study where the control group will receive the intervention after the intervention arm completes the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will be asked to complete Isha Kriya meditation twice daily for a total of six weeks in phase 1.
  Interventions: Behavioral: Isha Kriya Meditation
- Group 2 (Active Comparator): Participants will be asked to refrain from meditating for the first 6 weeks (phase 1) and then asked to complete Isha Kriya meditation for another 6 weeks (phase 2)
  Interventions: Behavioral: Isha Kriya Meditation

INTERVENTIONS:
Behavioral: Isha Kriya Meditation — Isha Kriya (IK) meditation is a meditation that can be learned quickly and requires approximately 12 minutes, twice a day practice. This regimen was chosen because it excels in simplicity and is a great way to introduce meditation to beginners. It does not incorporate a spiritual or religious focus. It was developed by the Isha Institute of Inner Sciences, a nonprofit foundation located at McMinnville, Tennessee.

SUMMARY:
This study will examine the effects of Isha Kriya meditation on stress and burnout among healthcare providers.

DETAILED DESCRIPTION:
In this study, investigators will evaluate the effect of Isha Kriya meditation on stress and burnout among perioperative healthcare providers. To do this, investigators will randomize healthy participants to one of two groups: one who will meditate twice daily for six weeks (group 1), and the other who will not meditate for first six weeks and then meditate for another six weeks (group 2). Investigators will then evaluate stress and burnout using validated electronic instruments at baseline and at six weeks for group 1 and at baseline, six weeks, and 12 weeks for group 2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Perioperative healthcare provider

Exclusion Criteria:

* Low English proficiency
* Currently enrolled in another interventional study that could impact the primary outcome, as determined by the Principal Investigator
* Not currently residing in the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in burnout levels among perioperative healthcare providers | From baseline to six weeks for group1 and baseline to 12 weeks for group 2
  Changes in burnout level due to meditation will be measured by Maslach Burnout Inventory (MBI)
Changes in stress levels among perioperative healthcare providers | From baseline to six weeks for group 1 and baseline to 12 weeks for group 2
  Changes in stress levels due to meditation will be measured by perceived stress scale (PSS; Scores can range from 0 to 40, with higher scores indicating higher perceived stress)
Changes in mood disturbances among perioperative healthcare providers | From baseline to six weeks for group 1 and baseline to 12 weeks for group 2
  Changes in mood disturbances due to meditation will be measured by profile of mood survey (POMS)

SECONDARY OUTCOMES:
Adherence to implementing a meditation program among healthcare providers. | From baseline to six weeks for group 1 and baseline to 12 weeks for group 2
  In this descriptive study, evaluation of feasibility will include adherence to meditation intervention (the proportion of completed meditation sessions out of the total required per protocol).

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided